CLINICAL TRIAL: NCT05709938
Title: Comparison of Insulin Glargine Mixed With Regular Insulin Versus the Standard Neutral Protamine Hagedorn (NPH) and Regular Insulin in the Treatment of Type 1 Diabetes Mellitus
Brief Title: Comparison of Insulin Glargine and Regular Insulin Versus NPH and Regular Insulin in the Treatment of T1DM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Glargine and regular insulin
Record Dates: First submitted 2023-01-14; First posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: To Assess the Glycemic Control of Insulin Glargine in Combination With Regular Insulin in Type 1 Diabetes in Children
MeSH Terms: interventions — Insulin Glargine; Insulin

STUDY DESIGN:
Intervention Model Description: 34 in each Arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Glargine (Experimental): Glargine-regular insulin regimen
  Interventions: Drug: Glargine and regular insulin versus NPH and regular insulin
- NPH (Active Comparator): NPH- regular insulin regimen
  Interventions: Drug: Glargine and regular insulin versus NPH and regular insulin

INTERVENTIONS:
Drug: Glargine and regular insulin versus NPH and regular insulin — Patients with type 1 diabetes (T1DM) in group A received insulin glargine as basal therapy at night and regular insulin given prior to each main meal.
  Patients in group B were given NPH and regular insulin in split and mix method in the morning and evening.

SUMMARY:
To compare the glycemic control in children with type 1 diabetes using insulin Glargine and regular insulin as basal bolus therapy versus Neutral Protamine Hagedorn insulin (NPH) and regular insulin.

DETAILED DESCRIPTION:
Diagnosed patients with Type-1 diabetes mellitus (T1DM), who had been on insulin therapy for more than three months, and met the eligibility criteria, were enrolled and randomly divided into group A and group B using the lottery method performed by the nursing staff.

Baseline HbA1c level was done for all the patients using CERA-STAT 2000 analyzer. The funding from KEMU was used to arrange insulin glargine and glucometer strips. The blood glucose levels of the patients were measured using the glucometer Freestyle Optium Neo H (manufactured by Abbott). Patients and their guardians were taught how to use the glucometer and record the measurements on monitoring sheets.

The total daily insulin dose was calculated according to the patient's age and pubertal stage for both groups. Patients in Group A (glargine-regular regimen) received insulin glargine (GLA) once in the evening (8:00 pm) and regular insulin 30 minutes before their three main meals. The starting dose of the GLA was 30% of the total daily insulin dose and titrated by 5-10 % according to the self-monitored fasting blood glucose levels to meet the age-appropriate goal range and avoid nocturnal hypoglycemia.

Patients in Group B (NPH-regular regimen) continued receiving NPH with regular insulin twice daily using the split and mix method, 30 minutes before breakfast and before dinner. NPH comprised 70% of the total daily dose. NPH titration was similar to that of the GLA group.

Each patient measured their capillary blood glucose levels 4-6 times per day as follows: pre-breakfast and 2-hours after breakfast, pre-lunch and 2-hours after lunch, pre-dinner and 2-hours after dinner. This monitoring continued for 90 days of the trial period.

Mid-night glucose levels were checked once weekly between 12 am and 3 am to check for hypolycemia or hyperglycemia, and that gave us 12 readings for the 90 days trial.

Each monitoring sheet presented the readings of pre-meals and 2-hours-post meals capillary blood glucose levels for each patient for 30 days. (annexure-B) All patients were followed up fortnightly at the Pediatric endocrine and diabetes section, Pediatric department, Mayo Hospital. Patients' compliance, insulin administration, and storage were assessed on each visit by asking the patient and the guardian. If needed, they were taught by the doctor and nurse attending the clinic. Both groups were instructed to walk daily for 20- 30 minutes and have three main meals and three snacks with avoidance of high carbohydrate dietary items. The patients had to mark their compliance with the instructed exercise and diet plan in the monitoring sheets.

The monitoring sheets were collected monthly during the study trial. After 90 days of the study, their HbA1C levels were tested using the same analyzer mentioned above for the baseline HbA1c.

ELIGIBILITY:
Inclusion Criteria:

* Children of age 3 to 18 years with Type 1 Diabetes Mellitus

Exclusion Criteria:

* Children below or above 18 years
* Comorbidities like celiac disease, hypothyroidism

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
HbA1c | Three months
  Baseline HbA1c is compared with the end HbA1c after 3 months of therapy
Hypoglycemia | Three months
  Capillary blood sugar level below 70mg/dl
Fasting blood sugar | Three months
  Capillary blood sugar before breakfast
Post-meal blood | Three months
  Capillary blood sugar level 2 hours after the three main meals
Mid night blood glucose level | Three months
  Capillary blood glucose levels between 12:00am -3:00am

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric endocrine and diabetes section, Pediatric department, Mayo Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Kliegman R, Stanton B, Geme J, Schor, Behrman R editor. Nelson textbook of pediatrics.20th ed. Canada: Elsevier; 2015.2763-2783.
- [Background] 2. American Diabetes Association. 2. Classification and diagnosis of diabetes: standards of medical care in diabetes-2018. Diabetes care. 2018 Jan 1;41(Supplement 1):S13-27.
- [Background] Aziz KM. Management of type-1 and type-2 diabetes by insulin injections in diabetology clinics - a scientific research review. Recent Pat Endocr Metab Immune Drug Discov. 2012 May;6(2):148-70. doi: 10.2174/187221412800604608. PMID 22559241
- [Background] Cryer P. Hypoglycemia in diabetes: pathophysiology, prevalence, and prevention. American Diabetes Association; 2016 Jul 12.
- [Background] Oyer DS. The science of hypoglycemia in patients with diabetes. Curr Diabetes Rev. 2013 May;9(3):195-208. doi: 10.2174/15733998113099990059. PMID 23506375
- [Background] Marra LP, Araujo VE, Silva TB, Diniz LM, Guerra Junior AA, Acurcio FA, Godman B, Alvares J. Clinical Effectiveness and Safety of Analog Glargine in Type 1 Diabetes: A Systematic Review and Meta-Analysis. Diabetes Ther. 2016 Jun;7(2):241-58. doi: 10.1007/s13300-016-0166-y. Epub 2016 Apr 5. PMID 27048292
- [Background] Hassan K, Rodriguez LM, Johnson SE, Tadlock S, Heptulla RA. A randomized, controlled trial comparing twice-a-day insulin glargine mixed with rapid-acting insulin analogs versus standard neutral protamine Hagedorn (NPH) therapy in newly diagnosed type 1 diabetes. Pediatrics. 2008 Mar;121(3):e466-72. doi: 10.1542/peds.2007-1679. Epub 2008 Feb 25. PMID 18299307
- [Background] Liu M, Zhou Z, Yan J, Li P, Song W, Fu J, Chen X, Zhao W, Xi L, Luo X, Sha L, Deng X, Gong C. A randomised, open-labelstudy of insulin glargine or neutral protamine Hagedorn insulin in Chinese paediatric patients with type 1 diabetes mellitus. BMC Endocr Disord. 2016 Nov 26;16(1):67. doi: 10.1186/s12902-016-0146-2. PMID 27887605
- [Background] Rostami P Md, Setoodeh A Md, Rabbani A Md, Nakhaei-Moghadam M Md, Najmi-Varzaneh F Md, Rezaei N Md PhD. A Randomized Clinical Trial of Insulin Glargine and Aspart, Compared to NPH and Regular Insulin in Children with Type 1 Diabetes Mellitus. Iran J Pediatr. 2014 Apr;24(2):173-8. PMID 25535536
- [Background] Tricco AC, Ashoor HM, Antony J, Beyene J, Veroniki AA, Isaranuwatchai W, Harrington A, Wilson C, Tsouros S, Soobiah C, Yu CH, Hutton B, Hoch JS, Hemmelgarn BR, Moher D, Majumdar SR, Straus SE. Safety, effectiveness, and cost effectiveness of long acting versus intermediate acting insulin for patients with type 1 diabetes: systematic review and network meta-analysis. BMJ. 2014 Oct 1;349:g5459. doi: 10.1136/bmj.g5459. PMID 25274009